CLINICAL TRIAL: NCT01446393
Title: Functional and Structural Characterization of the Peripheral Arteriopathy in Pseudoxanthoma Elasticum (PXE)
Brief Title: Functional and Structural Characterization of Arteriopathy in Pseudoxanthoma Elasticum (PXE)
Acronym: Ca-Art-PXE
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: CHU-Promoteur 2010-01
Record Dates: First submitted 2011-10-03; First posted 2011-10-05 (Estimated); Last update posted 2012-11-15 (Estimated); Status verified 2012-11

CONDITIONS: Pseudoxanthoma Elasticum
MeSH Terms: conditions — Pseudoxanthoma Elasticum

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples for genetic and serum analysis
Oversight: Data Monitoring Committee: No

SUMMARY:
To determine the specific structural and functional features of the peripheral arteriopathy in the Pseudoxanthoma Elasticum (PXE), an inherited autosomal disease.

DETAILED DESCRIPTION:
The primary objective of this study is to characterize the structural and functional characteristics of the peripheral arteries (lower and upper limbs) . a secondary objective will be to determine the arterial calcification using CT-scan as a useful tools for the diagnosis and the follow-up of this disease. Data will be collected from a cohort of patients PXE monitored in our Health and Research PXE center at the University Hospital of Angers. The structural and functional variables of the distal arteries (radial and tibialis arteries) will be studied using high-resolution echography. Scoring of the arterial calcium load will be determined by helicoidal CT-scan in the lower limb arteries. These variables will be compared to matched (gender and age) controls without PXE.

ELIGIBILITY:
Inclusion Criteria:

* Patients with phenotypically and genetically (ABCC6) proved PXE or control patients paired for age and gender
* Written formed consent obtained
* Patient affiliated to a Health care system

Exclusion Criteria:

* Patient with unproved PXE
* Pregnant woman
* Patient unwilling to participate to the study
* Not affiliated to a Health care System

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with phenotypically and genetically (ABCC6) proved PXE and Control patients paired for age (+/- 5 yeas) and gender.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2010-05; Primary Completion 2011-05 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Ludovic, MD, PhD, Principal Investigator — Department of Dermatology, University Hospital of Angers, France
Locations (1):
- Ludovic MARTIN, Angers, Pays de Loire, France

REFERENCES:
- [Background] Naouri M, Boisseau C, Bonicel P, Daudon P, Bonneau D, Chassaing N, Martin L. Manifestations of pseudoxanthoma elasticum in childhood. Br J Dermatol. 2009 Sep;161(3):635-9. doi: 10.1111/j.1365-2133.2009.09298.x. Epub 2009 Jun 9. PMID 19519828
- [Background] Martin L, Maitre F, Bonicel P, Daudon P, Verny C, Bonneau D, Le Saux O, Chassaing N. Heterozygosity for a single mutation in the ABCC6 gene may closely mimic PXE: consequences of this phenotype overlap for the definition of PXE. Arch Dermatol. 2008 Mar;144(3):301-6. doi: 10.1001/archderm.144.3.301. PMID 18347285
- [Derived] Martin L, Hoppe E, Kauffenstein G, Omarjee L, Navasiolava N, Henni S, Willoteaux S, Leftheriotis G. Early arterial calcification does not correlate with bone loss in pseudoxanthoma elasticum. Bone. 2017 Oct;103:88-92. doi: 10.1016/j.bone.2017.06.017. Epub 2017 Jun 27. PMID 28658601